CLINICAL TRIAL: NCT06228495
Title: Recovery at Your Fingertips: Pilot Study of an mHealth Intervention for Work-Related Stress Among Nursing Students (DIARY)
Brief Title: mHealth Intervention for Work-Related Stress
Acronym: DIARY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Aleksandra Sjöström-Bujacz, Assistant Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SFO-V 2021-2022 ASB
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Work Related Stress
Keywords: work stress; work-related stress; occupational stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Support (Experimental): This version of the intervention prompted users to engage in social support which is thought to buffer against the negative effects of stress. This effect is present in occupational settings, with several studies indicating that social support plays an important role in preventing burnout among nurses. Furthermore, interventions targeting social support in the workplace suggest that these have positive effects on mental health. Sample strategies included asking for help from co-workers, listening with compassion, and sharing authentic emotions.
  Interventions: Behavioral: Daily Intervention for Active Recovery
- Physical Activity (Active Comparator): This version of the interventions promoted an increase of physical activity in daily life. Physical activity is well-known to improve various health outcomes similar to our outcomes of interest, for instance reducing stress and burnout symptoms. Additionally, physical activity interventions in the workplace are widely used and have been found effective in many studies. Sample strategies included taking walks, going to the gym, and using the stairs instead of the elevator.
  Interventions: Behavioral: Daily Intervention for Active Recovery
- Psychological Strategies (Active Comparator): This version of the intervention promoted a variety of psychological strategies for stress reduction. Sample strategies included sleep quality improvement tips, mindfulness, and work detachment - evidence-based strategies that have a positive effect on outcomes of interest. Workplace interventions targeting these kinds of strategies have been found to be effective.
  Interventions: Behavioral: Daily Intervention for Active Recovery

INTERVENTIONS:
Behavioral: Daily Intervention for Active Recovery — Daily Intervention for Active Recovery - DIARY - is a 28-day intervention during which participants are prompted once daily to engage with intervention content. Each daily intervention interaction includes a short questionnaire with questions regarding sleep quality, current mood (e.g., tense, relaxed), and energy levels. Participants were prompted to open the application through a notification at 18:00 each evening. In case they did not fill out the questionnaire, an additional reminder notification was sent out at 20:00. The questionnaire closed each night at 03:00 am, at which point it was no longer possible to access the questionnaire for that day. The questionnaire took at most 5 minutes to complete. Upon completing the daily questionnaire participants received a prompt - a "bit-size" amount of information regarding stress and recovery as well as suggestions for a specific recovery strategy.

SUMMARY:
The objective of the trial is to pilot test the study protocol of a preventive, low-intensive mobile health (mHealth) intervention for work-related stress among nursing students. Work stress is a wide-spread problem affecting individual health as well as incurring substantial societal costs. mHealth solutions are among the most promising options for providing effective, scalable, and standardized interventions to employees.

DETAILED DESCRIPTION:
Researchers generally agree that recovery is a key buffer against the negative consequences of stress. Recovery behaviors, such as mindfulness and physical activity, are well-known to have a positive effect on stress-related health problems. For this reason, a behavior change intervention that successfully improves recovery may be effective in combating the long-term effects of stress. In this pilot study, three groups of participants received different versions of an intervention, each version containing a distinct set of recovery strategies.

The motivation of the present study is to pilot test the intervention and a study protocol in preparation for a future randomized controlled trial (RCT). Pilot testing the intervention and study procedures at an early stage is critical to identify potential pitfalls that need to be addressed before conducting a full-scale trial. Through investigating the study and intervention in preparatory phases we can refine the study protocol and intervention design in order to maximize the chances of a successful RCT.

The research questions for this pilot study are:

1. Data collection procedure - What is the recruitment and retention rate of invited participants? Does the randomization algorithm function properly?
2. Engagement - How often do participants use the intervention? Do they find the application easy and engaging to use?
3. Acceptability - Do participants find the intervention overall satisfactory and perceive it as beneficial? Is the digital tool technically stable?
4. Measurement quality - What is the completion rate for questionnaire items? What is the within-person variability in the daily measures?

ELIGIBILITY:
Inclusion Criteria:

* Active employee or student.

Exclusion Criteria:

* No psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Adherence | Over the course of the 28-day intervention.
  Adherence was operationalized as a count variable coded 0-28 representing the number of days that a given participant used the intervention.
App Engagement | At post-intervention, immediately after finishing the 28-day intervention.
  App Engagement was measured using The App Engagement Scale, a 7-item questionnaire designed to measure engagement with mobile applications, translated into Swedish by the research team. This translation has been used previously by the research team and has preliminary evidence of good reliability. Items (e.g. "I enjoyed using the app") are scored on a 1-5 ordered categories scale (1 = Not at all, 5 = Fully agree).
Daily stress | This was measured at once daily during the course of the 28-day intervention.
  Stress was measured daily as the mean value of three items inspired by the Stress-Energy Questionnaire. This study used a Swedish translation which has been validated in a previous study by the research team. Items ("During the last day, to what extent have you felt tense / pressed / frustrated?") were rated on a 6-point ordered categories scale (1 = Not at all, 6 = Very much). This variable was measured daily during the intervention and was not included in the pre-, post-, and follow-up measures.
Acceptability | At post-intervention, immediately after finishing the 28-day intervention.
  Acceptability was measured using a set of single-item measures evaluating whether the intervention was relevant to the user, if they would like to use it again, quality of the prompts, and technical stability. These items were only included in the post-intervention measure.

SECONDARY OUTCOMES:
Change in anxiety as measured by the Generalized Anxiety Disorder 7-item scale between baseline and post and follow-up measures. | This was measured at three time-points separated by one month each - baseline, post-intervention, follow-up.
  Anxiety was measured using the GAD-7 questionnaire, a 7-item instrument designed to assess generalized anxiety disorder. This study uses a Swedish translation. Items (e.g. "Feeling nervous, anxious, or on edge") were scored on a 1-4 ordered categories scale (1 = Not at all, 4 = Nearly every day).
Change in mindfulness as measured by the Mindful Attention Awareness Scale between baseline, post and follow-up measures. | This was measured at three time-points separated by one month each - baseline, post-intervention, follow-up.
  Mindfulness was measured using the Mindful Attention Awareness Scale, a 15-item measure designed to assess attention and awareness of "what is occurring in the present moment". This study used a Swedish translation with six items centered around emotional self-awareness. Items ("I could be experiencing some emotion and not be conscious of it until some time later") are rated on a 1-7 ordered categories scale (1 = Almost never, 7 = Almost always).
Change in recovery experiences as measured by the Recovery Experience Questionnaire between baseline, post and follow-up measures. | This was measured at three time-points separated by one month each - baseline, post-intervention, follow-up.
  Recovery was measured using the Recovery Experience Questionnaire, a 16-item questionnaire designed to measure four dimensions of recovery - detachment, relaxation, autonomy, and mastery - using four items for each dimension. This study uses a Swedish translation. Items ("In my free time I don't think about work") are scored on a 1-7 ordered categories scale (1 = Almost never, 7 = Almost always).
Change in exhaustion and disengagement from work as measured by the Oldenburg Burnout Questionnaire between baseline and post and follow-up measures. | This was measured at three time-points separated by one month each - baseline, post-intervention, follow-up.
  Exhaustion and disengagement from work was measured using the Oldenburg Burnout Inventory, an instrument designed to measure burnout in an occupational context including the dimensions exhaustion and disengagement. This study used a Swedish translation with a subset of 7 items. Items (e.g. "after work I often feel tired and exhausted") are scored on a 4-point ordered categories scale (1 = Not at all, 4 = Exactly).
Change in emotional exhaustion as measured by the Shirom-Melamed Burnout Questionnaire between baseline and post and follow-up measures. | This was measured at three time-points separated by one month each - baseline, post-intervention, follow-up.
  Emotional exhaustion was measured using the Shirom-Melamed Burnout Questionnaire (SMBQ), an instrument designed to assess burnout symptoms. The study used a Swedish translation and subset of 6 items focused on the emotional exhaustion dimension of burnout. Items ("My batteries are empty") are rated on a 1-7 ordered categories scale (1 = Almost never, 7 = Almost always).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Sjöström-Bujacz, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadzibajramovic E, Ahlborg G Jr, Grimby-Ekman A, Lundgren-Nilsson A. Internal construct validity of the stress-energy questionnaire in a working population, a cohort study. BMC Public Health. 2015 Feb 25;15:180. doi: 10.1186/s12889-015-1524-9. PMID 25885917
- [Background] Hansen E, Lundh LG, Homman A, Wangby-Lundh M. Measuring mindfulness: pilot studies with the Swedish versions of the Mindful Attention Awareness Scale and the Kentucky Inventory of Mindfulness Skills. Cogn Behav Ther. 2009;38(1):2-15. doi: 10.1080/16506070802383230. PMID 19125361
- [Background] Johansson R, Carlbring P, Heedman A, Paxling B, Andersson G. Depression, anxiety and their comorbidity in the Swedish general population: point prevalence and the effect on health-related quality of life. PeerJ. 2013 Jul 9;1:e98. doi: 10.7717/peerj.98. Print 2013. PMID 23862109
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sundstrom A, Soderholm A, Nordin M, Nordin S. Construct validation and normative data for different versions of the Shirom-Melamed burnout questionnaire/measure in a Swedish population sample. Stress Health. 2023 Aug;39(3):499-515. doi: 10.1002/smi.3200. Epub 2022 Oct 1. PMID 36166816
- [Background] Lundgren-Nilsson A, Jonsdottir IH, Pallant J, Ahlborg G Jr. Internal construct validity of the Shirom-Melamed Burnout Questionnaire (SMBQ). BMC Public Health. 2012 Jan 3;12:1. doi: 10.1186/1471-2458-12-1. PMID 22214479
- [Background] Peterson U, Bergstrom G, Samuelsson M, Asberg M, Nygren A. Reflecting peer-support groups in the prevention of stress and burnout: randomized controlled trial. J Adv Nurs. 2008 Sep;63(5):506-16. doi: 10.1111/j.1365-2648.2008.04743.x. PMID 18727753
- [Background] Bakker D, Rickard N. Engagement in mobile phone app for self-monitoring of emotional wellbeing predicts changes in mental health: MoodPrism. J Affect Disord. 2018 Feb;227:432-442. doi: 10.1016/j.jad.2017.11.016. Epub 2017 Nov 9. PMID 29154165
- [Background] Vega-Escano J, Porcel-Galvez AM, Diego-Cordero R, Romero-Sanchez JM, Romero-Saldana M, Barrientos-Trigo S. Insomnia Interventions in the Workplace: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2020 Sep 2;17(17):6401. doi: 10.3390/ijerph17176401. PMID 32887475
- [Background] Karabinski T, Haun VC, Nubold A, Wendsche J, Wegge J. Interventions for improving psychological detachment from work: A meta-analysis. J Occup Health Psychol. 2021 Jun;26(3):224-242. doi: 10.1037/ocp0000280. PMID 34096763
- [Background] Conn VS, Hafdahl AR, Cooper PS, Brown LM, Lusk SL. Meta-analysis of workplace physical activity interventions. Am J Prev Med. 2009 Oct;37(4):330-9. doi: 10.1016/j.amepre.2009.06.008. PMID 19765506
- [Background] Hogan BE, Linden W, Najarian B. Social support interventions: do they work? Clin Psychol Rev. 2002 Apr;22(3):383-442. doi: 10.1016/s0272-7358(01)00102-7. PMID 17201192
- [Background] Velando-Soriano A, Ortega-Campos E, Gomez-Urquiza JL, Ramirez-Baena L, De La Fuente EI, Canadas-De La Fuente GA. Impact of social support in preventing burnout syndrome in nurses: A systematic review. Jpn J Nurs Sci. 2020 Jan;17(1):e12269. doi: 10.1111/jjns.12269. Epub 2019 Oct 15. PMID 31617309
- [Background] Naczenski LM, Vries JD, Hooff MLMV, Kompier MAJ. Systematic review of the association between physical activity and burnout. J Occup Health. 2017 Nov 25;59(6):477-494. doi: 10.1539/joh.17-0050-RA. Epub 2017 Oct 7. PMID 28993574
- [Background] Ozbay F, Johnson DC, Dimoulas E, Morgan CA, Charney D, Southwick S. Social support and resilience to stress: from neurobiology to clinical practice. Psychiatry (Edgmont). 2007 May;4(5):35-40. PMID 20806028